CLINICAL TRIAL: NCT04644185
Title: A Multicenter, Adaptive, Randomized, Double-blinded, Placebo-controlled Phase II/III Trial to Evaluate the Efficacy and Safety of Monoclonal Antibody SCTA01 Against SARS-CoV-2 in Hospitalized Patients With Severe COVID-19
Brief Title: The Efficacy and Safety of SCTA01 in Hospitalized Patients With Severe COVID-19
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Preclinical test showed reduced efficacy
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCTA01-B301
Record Dates: First submitted 2020-11-22; First posted 2020-11-25 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — upanovimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- SCTA01 Low Dose+BSC (Experimental): SCTA01in a lower dose+best supportive care
  Interventions: Drug: SCTA01
- SCTA01 High Dose+BSC (Experimental): SCTA01in a higher dose+best supportive care
  Interventions: Drug: SCTA01
- Placebo+BSC (Active Comparator): SCTA01 excipients+best supportive care
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SCTA01 — SCTA01, a recombinant anti-SARS-CoV-2 spike protein monoclonal antibody
  Other Names: Recombinant anti-SARS-CoV-2 spike protein monoclonal antibody
  Arms: SCTA01 High Dose+BSC; SCTA01 Low Dose+BSC
Other: Placebo — all SCTA01 excipients without active component+best supportive care
  Other Names: SCTA01 excipients
  Arms: Placebo+BSC

SUMMARY:
The study is a multicenter, adaptive, randomized, double-blinded and placebo-controlled Phase II/III trial, and will be conducted globally. The study is comprised of two parts: dose selection (Phase II) and pivotal treatment effect (Phase III).

DETAILED DESCRIPTION:
In this study, Phase II part will evaluate the efficacy, safety and PK of SCTA01 low dose+BSC, high dose+BSC and placebo+BSC in patients with severe COVID-19.

In Phase II part, subjects will be randomized at 1:1:1 ratio. At the end of Phase II part, a dose for the Phase III will be determined.

The Phase III part will evaluate the efficacy, safety, and immunogenicity of SCTA01 at the recommended dose recommended. Subjects in Phase III part will be randomized at 1:1 ratio to SCTA01+BSC and placebo+BSC groups.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with severe COVID-19 (5 point on NIH 8-point ordinal scale).
* Male or female adult ≥18 years of age at time of enrollment;
* Biological samples (not limited to any specific type) collected within 72 hours before randomization is laboratory-confirmed as SARS-CoV-2 infection (PCR or antigen-based diagnostic tests);
* ≤ 10 days since symptoms of COVID-19 onset.

Exclusion Criteria:

* Patients who need non-invasive ventilation or high flow oxygen (i.e., 6 point on the 8-point ordinal scale);
* Patients with critical COVID-19;
* Patients with Severe COVID-19 who received convalescent plasma or COVID-19 vaccine, or anti-SARS-CoV-2 spike (S) protein targeted therapy;
* Alanine-amino transferase (ALT) or aspartate transaminase (AST) is 5 times higher than the upper limit of the normal value;
* Estimated glomerular filtration rate (eGFR) <30 mL/min or on dialysis {eGFR calculated by Cockcroft-Gault formula (Cockcroft DW, 1976), Male: CrCL (mL/min) = [(140 - age) × weight (kg)] × 1/ [SCr (mg/dL) × 72]; Female: CrCL (mL/min) = [(140 - age) × weight (kg)] × 0.85/ [SCr (mg/dL) × 72]}.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-03-27 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2022-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhanghua Lan, PhD, Study Director — Sinocelltech Ltd.
Locations (7):
- SCT study site, Somers Point, New Jersey, United States
- SCT study site, Buenos Aires, Argentina
- SCT study site, Uberlândia, Brazil
- SCT study site, Talca, Chile
- SCT study site, Rionegro, Colombia
- SCT study site, Monterrey, Mexico
- SCT study site, Lima, Peru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Groups:
- Low dose group: SCTA01 15 mg/kg plus best supportive care (BSC)
- High dose group: SCTA01 50 mg/kg plus best supportive care (BSC)
- Placebo group: Placebo plus best supportive care (BSC)
Period: Overall Study
Arm/Group | Low dose group | High dose group | Placebo group
Started | 33 | 35 | 34
Completed | 33 | 35 | 34
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SCTA01 Low Dose+BSC | SCTA01 High Dose+BSC | Placebo+BSC | Total
Number analyzed (Participants) | 33 | 34 | 35 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 21 | 58
  >=65 years | 14 | 16 | 14 | 44
Age, Continuous [Median (Full Range); unit: years] | 48 [18 to 81] | 48 [30 to 69] | 44 [18 to 76] | 47 [18 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 10 | 34
  Male | 21 | 22 | 25 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 4 | 9
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 0 | 8
  White | 22 | 25 | 0 | 47
  More than one race | 0 | 0 | 29 | 29
  Unknown or Not Reported | 4 | 2 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Time to Clinical Improvement up to Day 29
Description: The median time to clinical improvement in the SCTA01 groups and control group
Time Frame: Day 29
Population: There is no difference beteeen the numbers of participants or units assigned to the arms or groups .
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Low dose group | High dose group | Placebo group
Number analyzed (Participants) | 33 | 34 | 35
days | 9 [7 to 14] | 9 [6 to 15] | 10 [7 to 15]

ADVERSE EVENTS:
Time Frame: The advese events were collected over 120 days
Description: An adverse event (AE) is any unfavorable or unintended sign, symptom, disease, or abnormal lab result related to a medicinal product, regardless of causality. It includes new/worsening conditions, procedure complications, lack of efficacy, overdose, misuse, or occupational exposure. A serious AE (SAE) results in death, life-threatening risk, hospitalization, disability, birth defect, or other important events.
Arm/Group | SCTA01 Low Dose+BSC | SCTA01 High Dose+BSC | Placebo+BSC
All-Cause Mortality (participants affected / at risk) | 2/33 | 2/34 | 3/35
Serious Adverse Events (participants affected / at risk) | 7/33 | 5/34 | 5/35
Other Adverse Events (participants affected / at risk) | 9/33 | 16/34 | 11/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCTA01 Low Dose+BSC (N=33) | SCTA01 High Dose+BSC (N=34) | Placebo+BSC (N=35)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Cardiac Disorder (Cardiac disorders) | 2 (2) | 1 (1) | 2 (2)
Infection (Infections and infestations) | 3 (3) | 3 (3) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCTA01 Low Dose+BSC (N=33) | SCTA01 High Dose+BSC (N=34) | Placebo+BSC (N=35)
Gastrointestinal disorders Constipaton (Gastrointestinal disorders) | 6 (6) | 11 (11) | 4 (4)
Pyrexia (General disorders) | 3 (3) | 6 (6) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 3 (3) | 4 (4)
Hypotension (Vascular disorders) | 1 (1) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/85/NCT04644185/Prot_SAP_000.pdf